CLINICAL TRIAL: NCT01113606
Title: A Double-Blind, Randomized, Controlled Trial to Assess the Effects of the Obagi Nu-Derm System on Re-Epithelialization After Chemical Peel or Ablative Laser Resurfacing.
Brief Title: A Trial of Skin Care Protocols for Facial Resurfacing
Acronym: SPAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Plastic Surgery Foundation (Other)
Other Study IDs: PSEF001-06
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Facial Photo Damage; Periocular Fine Wrinkles; Perioral Fine Wrinkles
Keywords: Moderate to severe facial photo damage; Periocular or perioral fine wrinkles
MeSH Terms: interventions — Standard of Care

ARMS (2):
- Obagi Nu-Derm System (ONDS) (Active Comparator)
  Interventions: Other: Obagi New-Derm System
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Obagi New-Derm System
  Arms: Obagi Nu-Derm System (ONDS)
Other: Standard of Care
  Arms: Standard of Care

SUMMARY:
The aims of the Skin Product Assessment Research study were to (1) develop an infrastructure and process for industry-sponsored, Plastic Surgery Educational Foundation (PSEF) research in facial aesthetic surgery and (2) test the research process by comparing outcomes of the Obagi Nu-Derm System (ODNS) and conventional therapy as treatment adjuncts in ablative facial resurfacing.

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate to severe photo damage and rhytids, undergoing full or partial face resurfacing with chemical peel or ablative laser.
* Fitzpatrick I-IV skin types

Exclusion Criteria:

* patients unable to complete the regimen or who had used topical prescription steroids, retinoids, depigmentation products or other products containing hydroquinone and polyhydroxy acids within 8 weeks of enrollment.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Suite 135, Oxnard, California
  - Suite 175, Rancho Santa Margarita, California
  - Aesthetic and Plastic Surgery Institute, Greeley, Colorado
  - Brevard Plastic Surgery and Skin Institute, Melbourne, Florida
  - Kentucky Aesthetic and Plastic Surgery Institute, Louisville, Kentucky
  - Center for Plastic and Reconstructive Surgery, Ypsilanti, Michigan
  - Body Aesthetic Plastic Surgery, St Louis, Missouri
  - New York, New York
  - Advanced Cosmetis Surgery, Greenville, South Carolina